CLINICAL TRIAL: NCT01171248
Title: Central and Peripheral 24h BP and the Association to Autonomic Neuropathy and Diabetic Nephropathy in Type 1 Diabetic Patients
Brief Title: Study of 24 Hour Blood Pressure and the Association to Complications to Type 1 Diabetes
Acronym: PROFIL
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Rossing, Senior Physician, DMSc, Steno Diabetes Center Copenhagen
Other Study IDs: PROFIL-H-B-2009-056
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Type 1 Diabetes; Hypertension
Keywords: nocturnal blood pressure dip; complications; ambulatory blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- type 1 diabetes
- non-diabetics

SUMMARY:
The aim of the study is to evaluate the prevalence of abnormal nocturnal blood pressure (BP) in patients with type 1 diabetes. The investigators wish to gain knowledge on the relation between central and peripheral 24 hour BP and a possible association to late complications in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* more than 18 years of age

Exclusion Criteria:

* End Stage Renal Disease (ESRD)
* dialysis
* other kidney disease than diabetic nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: type 1 diabetic patients (600 patients) non-diabetic controls (50)
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure (AMBP) | 2 years
  The participants are seen once (cross-sectional) and we measure AMBP in order for us to investigate any association between AMBP and other parameters such as age, duration of diabetes, albuminuria status and other diabetic complications.

SECONDARY OUTCOMES:
Diabetic late complications | 2 years
  The participants are only seen once and are at this visit, asked in regards to complications, and the electronic patient medical record is rewieved in regards to complications.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, MD, DmSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Hansen CS, Rasmussen DGK, Hansen TW, Nielsen SH, Theilade S, Karsdal MA, Genovese F, Rossing P. Collagen turnover is associated with cardiovascular autonomic and peripheral neuropathy in type 1 diabetes: novel pathophysiological mechanism? Cardiovasc Diabetol. 2023 Jun 29;22(1):158. doi: 10.1186/s12933-023-01891-8. PMID 37386485
- [Derived] Theilade S, Lajer M, Hansen TW, Rossing P. Pulse wave reflection is associated with diabetes duration, albuminuria and cardiovascular disease in type 1 diabetes. Acta Diabetol. 2014 Dec;51(6):973-80. doi: 10.1007/s00592-014-0651-6. Epub 2014 Oct 2. PMID 25274394
- [Derived] Theilade S, Lajer M, Hansen TW, Joergensen C, Persson F, Andresdottir G, Reinhard H, Nielsen SE, Lacy P, Williams B, Rossing P. 24-hour central aortic systolic pressure and 24-hour central pulse pressure are related to diabetic complications in type 1 diabetes - a cross-sectional study. Cardiovasc Diabetol. 2013 Aug 27;12:122. doi: 10.1186/1475-2840-12-122. PMID 23978271